CLINICAL TRIAL: NCT01827254
Title: Etude Resume (Retraitement Sunitinib Rein Metastatique)
Brief Title: Sutent Rechallenge In mRCC Patients
Acronym: RESUME
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181211; ETUDE RESUME (Other: Alias Study Number)
Record Dates: First submitted 2013-03-25; First posted 2013-04-09 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: sutent rechallenge
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-Interventional Study
  Interventions: Other: sunitinib: observational study

INTERVENTIONS:
Other: sunitinib: observational study — Observational study evaluating patients who were treated with sunitinib in 1st line and in 3rd line
  Other Names: sunitinib 50 mg 4/2

SUMMARY:
Retrospective and prospective study in mRCC patients treated with sutent in first line and rechallenged by Sutent in 3rd and 4th line.

DETAILED DESCRIPTION:
A sample size of n = 40 patients will allow to estimate of the median PFS with a precision around 1.8 months (based on data from Rini et al.) This retrospective and prospective study is designed to estimate the effect of Sutent rechallenge.

The PFS (estimated from Kaplan-Meier estimate) will be the primary endpoints. In addition, the effects of sunitinib at the 2 periods of treatment (i.e. first line sunitinib vs. rechallenge) will be compared by Wilcoxon signed-rank test for PFS values and by McNemar test for overall response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic RCC containing predominantly clear cell component.
* Previously received sunitinib in first line, 2 or more antitumor therapies subsequently and then received sunitinib for a second time.
* At least 1 cycle of sunitinib rechallenge (1 cycle= 4 weeks on/2 weeks off).
* At least 1 measurable lesion that can be accurately measured in at least 1 dimension with the longest diameter (LD) ³ 10 mm when measured by spiral computerized tomography (CT) (5-mm slice thickness contiguous) or ³ 20 mm when measured by conventional CT (10-mm slice thickness contiguous). The lesion must be ³ 2 times the size of the slice thickness per RECIST criteria.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Patient who didn't receive Sunitinib in first line.
* Patient who received less than one line of treatment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mRCC patients treated with sunitinib in first line and rechallenged with sunitinib in 3rd and 4th line
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- France (18):
  - CHU de la Timone, Marseille, Cedex 5
  - Hopital albert Michalon, Grenoble, Cedex 9
  - Departement d'Oncologie Medicale-Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez, France
  - Centre Paul Papin, Angers
  - Hôpital Saint-André, Bordeaux
  - Centre Catalan Urologie Andrologie, Cabestany
  - Centre Oscar Lambret - Cancérologie Urologie Digestive, Lille
  - clinique de la Louvière, Lille
  - Hopital Dupuytren - Oncologie Medicale, Limoges
  - Centre Leon Berard, Service d'Oncologie Medicale, Lyon
  - Institut Paoli-Calmettes / Hôpital de jour, Marseille
  - Hopital Timone Adultes, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Eugene Marquis, Rennes
  - CHU Charles Nicolle, Rouen
  - Centre Rene Gauducheau - Service Oncologie Medicale, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181211&StudyName=Sutent%20Rechallenge%20In%20mRCC%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who met the selection criteria and received first-line sunitinib as per standard local practice, followed by one or more lines of different treatments (bevacizumab with interferon, bevacizumab without interferon, sorafenib, axitinib, temsirolimus or everolimus), and, lastly were rechallenged with sunitinib between 2006 and May 2013 were included in this non-interventional study.
Period: Overall Study
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Started | 61
Evaluable Population | 52
Completed | 2
Not Completed | 59
Not completed — Death | 10
Not completed — Case report form not completed | 4
Not completed — Invalidated centre | 3
Not completed — Discontinued prior initiation: sunitinib | 1
Not completed — Did not complete re-challenge | 1
Not completed — Disease progression | 36
Not completed — Intolerance to treatment | 4

BASELINE CHARACTERISTICS:
Population: Evaluable population: All participants included in the analysis.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival With Sunitinib as First Line of Therapy
Description: The PFS was defined as the time interval between the start date of treatment and the date of progression as assessed by the investigator or date of death occurring after treatment initiation, whichever occurred first. Duration of progression free survival= [(Date of mRCC progression - Start date of the treatment) + 1)]/ 365.25 x 12. Progression was defined as an increase in visible disease.
Time Frame: From start of treatment up to 66.6 months
Population: Evaluable population: All participants included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with metastatic renal cell carcinoma (MRCC) who met the selection criteria and received sunitinib as first-line therapy as per standard local practice.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 52
months | 18.4 [12.5 to 23.7]

2. Secondary Outcome: Overall Survival
Description: Overall survival of patients under treatment was evaluated by calculating the time between date of initiation of treatment (1st line) and date of death, if the latter occurred before the end of the study. Duration of Overall Survival =(Date of death - Start date of treatment) + 1)/365.25 x 12.
Time Frame: Baseline up to death or end of study (up to 98.0 months)
Population: Evaluable population: All participants included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who met the selection criteria and received first-line sunitinib as per standard local practice, followed by one or more lines of different treatments (bevacizumab with interferon,bevacizumab without interferon, sorafenib,axitinib, temsirolimus or everolimus), and, lastly were rechallenged with sunitinib between 2006 and May 2013 were included in this non--interventional study.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 52
months | 55.9 [48.0 to 63.7]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target lesions and non-target lesions, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Percentage of participants with objective response was calculated for the 1st-line of therapy with Sunitinib, Sunitinib re-challenge and for retreatment with Sunitinib as 3rd-line of therapy or more.
Time Frame: Baseline up to 98.0 months
Population: Evaluable population: All participants included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 52
percentage of participants
  First line treatment | 53.8 [40.3 to 67.4]
  Third line treatment | 15.4 [5.6 to 25.2]
  Sunitinib re-challenge | 75.0 [45.0 to 100.0]

4. Other Pre Specified Outcome: Number of Participant With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs include both serious as well as non-serious AEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 24 months
Population: Evaluable population: All participants included in the analysis.
Measure: Number; unit: participants
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 52
participants
  AEs | 24 [48.0 to 63.7]
  SAEs | 21

5. Primary Outcome: Progression Free Survival for Re-challenge With Sunitinib
Description: as for outcome 1
Time Frame: From start of treatment up to 52.2 months
Population: Evaluable population: All participants included in the analysis. Here "N" signifies number of participants who were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who met the selection criteria and received first-line sunitinib as per standard local practice, followed by one or more lines of different treatments (bevacizumab with interferon,bevacizumab without interferon, sorafenib,axitinib, temsirolimus or everolimus), and, lastly were rechallenged with sunitinib between 2006 and May 2013 were included in this non-interventional study.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 51
months | 7.9 [5.4 to 13.2]

6. Primary Outcome: Progression Free Survival: Second Line of Treatment
Description: The PFS was defined as the time interval between the start date of treatment and the date of progression as assessed by the investigator or date of death occurring after treatment initiation, whichever occurred first. Duration of progression free survival= [(Date of mRCC progression - Start date of the treatment) + 1)]/ 365.25 x 12. Progression was defined as an increase in visible disease. Second-line treatment were divided in two groups: Group A (received treatment with: bevacizumab (with interferon), bevacizumab (without interferon), sorafenib, axitinib) and Group B (received treatment with: temsirolimus, everolimus).
Time Frame: From start of treatment up to 22.9 months
Population: Evaluable population: All participants included in the analysis. Here "N" signifies number of participants who were analyzed for this outcome measure and "n" signifies those participants who were evaluable for respective treatment group.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who met the selection criteria and received first-line sunitinib, followed by second line treatment with bevacizumab (with interferon),bevacizumab (without interferon), sorafenib, axitinib, temsirolimus or everolimus as per standard local practice.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 50
months
  Group A (n=21) | 5.0 [2.8 to 7.0]
  Group B (n=29) | 6.2 [3.7 to 7.9]

7. Primary Outcome: Progression Free Survival: Third Line Treatment
Description: The PFS was defined as the time interval between the start date of treatment and the date of progression as assessed by the investigator or date of death occurring after treatment initiation, whichever occurred first. Duration of progression free survival= [(Date of mRCC progression - Start date of the treatment) + 1)]/ 365.25 x 12. Progression was defined as an increase in visible disease. Third-line treatment were divided in two groups: Group A (received treatment with: bevacizumab (with interferon), bevacizumab (without interferon), sorafenib, axitinib) and Group B (received treatment with: temsirolimus, everolimus).
Time Frame: From start of treatment up to 23.7 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Renal Cell Carcinoma (mRCC) Cohort: Participants diagnosed with mRCC who met the selection criteria and received first-line sunitinib, followed by third line treatment with bevacizumab (with interferon), bevacizumab (without interferon), sorafenib, axitinib, temsirolimus or everolimus as per standard local practice.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Number analyzed (Participants) | 39
months
  Group A (n=20) | 4.8 [3.1 to 8.7]
  Group B (n=19) | 10.8 [7.0 to 14.6]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Metastatic Renal Cell Carcinoma (mRCC) Cohort
Serious Adverse Events (participants affected / at risk) | 21/52
Other Adverse Events (participants affected / at risk) | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Renal Cell Carcinoma (mRCC) Cohort (N=52)
Neutropenia (Blood and lymphatic system disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Disease progression (General disorders) | 9
General physical health deterioration (General disorders) | 2
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Confusional state (Psychiatric disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Renal Cell Carcinoma (mRCC) Cohort (N=52)
Anaemia (Blood and lymphatic system disorders) | 2
Macrocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Conjunctivitis (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 8
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Blood pressure inadequately controlled (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.